CLINICAL TRIAL: NCT07303270
Title: Assessing Emotional Processes in Adults With Intellectual Developmental Disorder Using the ACQUISS Battery
Brief Title: Emotional Processes in Adults With Intellectual Developmental Disorder
Acronym: EmoTDI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A01946-43
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Intellectual Developmental Disorder
Keywords: Intellectual Developmental Disorder; emotional processing; Cognitive assessments; Social cognition
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: IDD group compared to control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDD group (Experimental): adults with Intellectual Developmental Disorder
  Interventions: Other: ACQUISS protocol assessing emotional processing.
- Control group (Other): healthy adults
  Interventions: Other: ACQUISS protocol assessing emotional processing.

INTERVENTIONS:
Other: ACQUISS protocol assessing emotional processing. — Task 1: 5 minute facial emotion recognition test to identify isolated facial expressions. 6 drawn faces, without gender bias, without hair, expressing the 6 universal emotions will be presented. The emotions are: happiness, sadness, anger, fear, surprise and disgust.
  Task 2 : identifying a character's emotion in a social context (20 min). The subject is presented with drawn social contexts, one character is always in orange, and the face is left blank. The subject then has to choose amongst 6 emotions (happiness, sadness, anger, fear, surprise and disgust) which one would correspond the most to the emotion expressed by the character in orange.
  Task 3 : recognizing vocal emotions (15 min). The subject is presented with dialogues of 3 sentences. The 3 sentences are expressed with a vocal emotion (same emotion for the 3 sentences). The contents of the sentences are neutral At the end of each dialogue, the subject has to show which emotion was expressed.

SUMMARY:
Emotions play a crucial part in the quality of life, interpersonal relationships and mental health in general. In adults presenting with intellectual developmental disorder (IDD), emotional abilities may be hindered, thus leading to more challenging behaviors. A better understanding of emotional processes of adults with IDD may help improve the efficiency of behavioral interventions and better improve their quality of life.

The primary goal of this study is to better characterize the abilities and weaknesses of adults with IDD concerning their emotional processes, in comparison to a healthy population. The secondary goals are :

* to determine if these difficulties are underlined by oculomotor and attention (auditory and visual) processes
* to determine if behavioral difficulties, as reported by the families of adults with IDD, are underlined by specific difficulties in facial emotion recognition, emotion identification in context and/or identification of vocal emotions.

DETAILED DESCRIPTION:
The study will be carried out in 3 steps :

Step 1: All participants will undergo tests to evaluate their intellectual abilities, and auditory and visual screening tests.

Step 2 : All participants will undergo neuropsychological tests assessing attentional and oculomotor abilities (1 hour). During this time, the participant's family member will complete the questionnaires assessing behavior.

Step 3 : All participants will undergo the experimental ACQUISS protocol (task 1 : faces; task 2 : faces in context; task 3 : prosody) (1 hour).

Detailed Description:

Step 1 :

During this first step, all participants (both groups), will undergo the Raven Progressive Matrices (John and Raven 2003) to assess their intellectual abilities. They will then undergo an auditory screening test (tonality test) and a visual screening task (the Rossano-Weiss scale and the Palettes de Léa Grattins task).

Step 2 :

During this second step, all participants (both groups) will undergo :

1. - the tangled lines test (Rey, 1964) : in this task, the participant must follow by gaze entangled lines to determine the beginning and end of each line.
2. - the NSUCO oculomotor test (Maillet, 2015) : the orthoptist will evaluate the ability of the participant to carry out ocular saccades and movement pursuit.
3. - the Auditory attention task of the NEPSY-II battery (Korkman et al., 2012)
4. - 2 cancellation tests from the EVA battery (Chokron, 2010):

   * the TeddyBear Cancellation test
   * the single-letter cancellation test

Step 3:

During this step, all participants from both groups will undergo the ACQUISS protocol.

ELIGIBILITY:
Inclusion Criteria:

IDD group :

* Diagnosis of IDD according to DSM-V criteria
* aged between 18 and 3 years
* French speaking
* Membership or entitlement to a social security plan
* informed consent, or that of the tutor, to take part in the study
* presence of a caregiver to complete the questionnaires at V2.

Control group :

* aged between 18 and 35 years
* French speaking
* Membership or entitlement to a social security plan
* Informed written consent to take part in the study.

Exclusion Criteria:

IDD group :

* visual or auditory impairments, evaluated at V1
* non stabilized epilepsy
* undergoing treatments that can impact brain or psychological functioning
* major motor disorders
* breastfeeding or pregnant woman

Control group :

* neurodevelopmental or psychiatric disorder
* history of brain trauma (TBI, stroke, etc…) or non-stabilized epilepsy
* visual or auditory impairments, evaluated at V1
* non stabilized epilepsy
* undergoing treatments that can impact brain or psychological functioning
* major motor disorders
* breastfeeding or pregnant woman

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-07-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
proportion of correct answers on the ACQUISS battery | Baseline
  proportion of correct answers in each of the 3 tasks

SECONDARY OUTCOMES:
Proportion of correct answers on the Entangled lines test | Baseline
Proportion of correct answers on the NSUCO test | Baseline
  Northeastern State University College of Optometry test.
Proportion of correct answers on an auditory attentional task (NEPSY-II) | Baseline
Proportion of correct signs barred on the TeddyBear task | Baseline
Proportion of correct signs barred on the letter task | Baseline
Score on the Agressivity questionnaire | Baseline
  Score on the Agressivity questionnaire ("Problematic behavior in group settings"), filled in by a caregiver. Minimum score = 6; Maximum score = 30. Higher scores suggest greater agressivity.
Score on the Aberrant Behavior Checklist | Baseline
  Score on the Aberrant Behavior Checklist, filled in by a caregiver. Minimum = 0; Maximum = 174. Higher scores reflect more severe levels of challenging behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- CH Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided